CLINICAL TRIAL: NCT00917579
Title: An Open Label, Randomized, Single Dose, Two-Way Crossover Bioequivalence Study Comparing A New 10 Mg Atorvastatin Tablet To A 10 Mg Atorvastatin Commercial Tablet In Healthy Subjects
Brief Title: Bioequivalence Study Comparing A New 10 Mg Atorvastatin Tablet To A 10 Mg Atorvastatin Commercial Tablet
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: A2581166
Record Dates: First submitted 2009-06-08; First posted 2009-06-10 (Estimated); Results first posted 2009-10-14 (Estimated); Last update posted 2021-03-12 (Actual); Status verified 2021-02

CONDITIONS: Hypercholesterolemia
Keywords: Bioequivalence, pharmacokinetics, atorvastatin
MeSH Terms: conditions — Hypercholesterolemia | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reference (Other): 10 mg atorvastatin
  Interventions: Drug: Atorvastatin
- Test (Experimental): New 10 mg atorvastatin tablet
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — A single 10 mg dose of marketed 10 mg atorvastatin tablets
  Arms: Reference
Drug: Atorvastatin — A single 10 mg dose of new formulation of 10 mg atorvastatin
  Arms: Test

SUMMARY:
• To determine whether new 10 mg atorvastatin tablets are bioequivalent to 10 mg commercial atorvastatin tablets (Lipitor®).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 18 and 55 years
* Body Mass Index (BMI) of 18 to 30 kg/m2; and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing) disease or clinical findings at screening.
* Treatment with an investigational drug within 30 days or 5 half lives preceding the first dose of study medication.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2008-07; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Miami, Florida, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A2581166&StudyName=Bioequivalence%20Study%20Comparing%20A%20New%2010%20Mg%20Atorvastatin%20Tablet%20To%20A%2010%20Mg%20Atorvastatin%20Commercial%20Tablet

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy volunteers were recruited from one research center between July 2008 and September 2008.
Groups:
- Test Drug First, Then Reference Drug: New (test) 10 milligram (mg) atorvastatin tablet as a single oral dose in the first intervention period, and marketed (reference) 10 mg atorvastatin tablet as a single oral dose in the second intervention period (after washout period).
- Reference Drug First, Then Test Drug: Marketed (reference) 10 mg atorvastatin commercial tablet (Lipitor®) as a single oral dose in the first intervention period, and new (test) 10 mg atorvastatin tablet as a single oral dose in the second intervention period (after washout period).
Period: Period 1: 1st Intervention
Arm/Group | Test Drug First, Then Reference Drug | Reference Drug First, Then Test Drug
Started | 39 | 37
Completed | 39 | 37
Not Completed | 0 | 0
Period: Washout >= 2 Weeks
Arm/Group | Test Drug First, Then Reference Drug | Reference Drug First, Then Test Drug
Started | 39 | 37
Completed | 37 | 37
Not Completed | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Period 2: 2nd Intervention
Arm/Group | Test Drug First, Then Reference Drug | Reference Drug First, Then Test Drug
Started | 37 | 37
Completed | 37 | 37
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total Number of Participants: All participants received atorvastatin 10 mg tablets (new and marketed).
Arm/Group | Total Number of Participants
Number analyzed (Participants) | 76
Age, Customized [Number; unit: participants]
  18-44 years | 59
  45-64 years | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 38

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUC Infinity)
Description: AUCinf = Area under the plasma concentration-time curve from time 0 (predose) extrapolated to infinite time; measured in nanograms times hour per milliliter (ng•hr/mL).
Time Frame: 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 10, 12, 24, 36, 48, 72 hours post dose
Population: Pharmacokinetic (PK) parameter analysis population: all subjects enrolled and treated who had at least 1 of the PK parameters of primary interest in at least 1 treatment period. Only 73 subjects contributed to the PK analysis in the reference group as plasma concentrations for 1 subject were below the limit of quantification, except 1 time point.
Measure: Mean (Standard Deviation); unit: ng•hr/mL
Groups:
- Test Drug: New (test) 10 mg atorvastatin tablet as a single oral dose in either first intervention period or second intervention period.
- Reference Drug: Marketed (reference) 10 mg atorvastatin tablet (Lipitor®) as a single oral dose in either first intervention period or second intervention period.
Arm/Group | Test Drug | Reference Drug
Number analyzed (Participants) | 76 | 73
ng•hr/mL | 18.3206 (8.26454) | 19.2583 (8.79739)
Statistical Analysis 1: Comparison: Test Drug vs Reference Drug; Natural log transformed AUCinf was analyzed using a mixed effects model with sequence, period and treatment as fixed effects and subject within sequence as a random effect. Adjusted mean difference (Test-Ref) and 90% CI was obtained from the model and exponentiated to provide estimates of the ratio of adjusted geometric mean and 90% CI for the ratio. Alternative hypothesis of bioequivalence: (H1: θL <=µT - µR <=θU); null hypothesis of inequivalence: (Ho: µT - µR <θL or µT - µR >θU); Test type: Non-Inferiority or Equivalence — Bioequivalence of the two treatments was concluded if the 90% confidence intervals for the ratio of adjusted geometric means for both AUCinf and Cmax fell within (80%, 125%); ANOVA; Values were back-transformed from the log scale; ratio of adjusted geometric means = 95.34, 90% CI [91.33 to 99.52] — Parameter estimate = ratio (%) (test/reference) of adjusted geometric means. AUClast + (Clast*/kel), where Clast* was the predicted plasma concentration at the last quantifiable time point estimated from the log-linear regression analysis

2. Primary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast)
Description: AUClast = area under the plasma concentration-time curve from 0 (predose) to the time of the last measureable concentration (Clast); measured in nanograms times hour per milliliter (ng•hr/mL).
Time Frame: 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 10, 12, 24, 36, 48, 72 hours post dose
Population: PK parameter analysis population: all subjects enrolled and treated who had at least 1 of the PK parameters of primary interest in at least 1 treatment period. Only 73 subjects contributed to the PK analysis in the reference group as plasma concentrations for 1 subject were below the limit of quantification, with the exception of 1 time point.
Measure: Mean (Standard Deviation); unit: ng•hr/mL
Arm/Group | Test Drug | Reference Drug
Number analyzed (Participants) | 76 | 73
ng•hr/mL | 15.7382 (7.88920) | 16.5452 (8.71551)
Statistical Analysis 1: Comparison: Test Drug vs Reference Drug; Natural log transformed AUClast was analyzed using a mixed effects model with sequence, period and treatment as fixed effects and subject within sequence as a random effect. Estimates of the adjusted mean differences (Test-Reference) and corresponding 90% confidence interval was obtained from the model and exponentiated to provide estimates of the ratio of adjusted geometric mean (Test/Reference) and 90% confidence interval for the ratio; Test type: Non-Inferiority or Equivalence — Bioequivalence of the two treatments was concluded if the 90% confidence intervals for the ratio of adjusted geometric means for both the AUCinf and Cmax fell within (80%, 125%). AUCinf method of determination includes AUC last calculated value; ANOVA; Values have been back-transformed from the log scale; ratio of adjusted geometric means = 95.79, 90% CI [91.07 to 100.76] — Parameter estimate = ratio (%) (test/reference) of adjusted geometric means. Log-linear trapezoidal method

3. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Description: Cmax = maximum observed plasma concentration. Measured in nanograms per milliter (ng/mL).
Time Frame: 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 10, 12, 24, 36, 48, 72 hours post dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Test Drug | Reference Drug
Number analyzed (Participants) | 76 | 73
ng/mL | 2.6594 (1.44617) | 2.8086 (1.23048)
Statistical Analysis 1: Comparison: Test Drug vs Reference Drug; Natural log transformed Cmax was analyzed using a mixed effects model with sequence, period and treatment as fixed effects and subject within sequence as a random effect. Estimates of the adjusted mean differences (Test-Reference) and corresponding 90% confidence intervals were obtained from the model and exponentiated to provide estimates of the ratio of adjusted geometric mean (Test/Reference) and 90% confidence interval for the ratio; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Values have been back-transformed from the log scale; ratio of adjusted geometric means = 91.41, 90% CI [83.39 to 100.20] — Parameter estimate = ratio (%) (test/reference) of adjusted geometric means

4. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax)
Description: Tmax = time (hours) to maximum plasma concentration (Cmax).
Time Frame: 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 10, 12, 24, 36, 48, 72 hours post dose
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Test Drug | Reference Drug
Number analyzed (Participants) | 76 | 73
hours | 1.000 [0.250 to 9.000] | 0.5000 [0.250 to 4.000]

5. Secondary Outcome: Plasma Elimination Half-life (t1/2)
Description: t1/2 = terminal elimination half-life in hours.
Time Frame: 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 10, 12, 24, 36, 48, 72 hours post dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Test Drug | Reference Drug
Number analyzed (Participants) | 76 | 73
hours | 10.39 (4.0018) | 10.78 (3.9640)

ADVERSE EVENTS:
Groups:
- Test Drug: New (test) 10 mg atorvastatin tablet as a single oral dose.
- Reference Drug: Marketed (reference) 10 mg atorvastatin tablet (Lipitor®) as a single dose.
Arm/Group | Test Drug | Reference Drug
Serious Adverse Events (participants affected / at risk) | 1 | 0
Other Adverse Events (participants affected / at risk) | 4 | 15
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Test Drug | Reference Drug
Renal colic (Renal and urinary disorders) | 1/76 | 0/74
OTHER ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Test Drug | Reference Drug
Constipation (Gastrointestinal disorders) | 1/76 | 4/74
Dyspepsia (Gastrointestinal disorders) | 0/76 | 1/74
Nausea (Gastrointestinal disorders) | 0/76 | 2/74
Vomiting (Gastrointestinal disorders) | 0/76 | 1/74
Dizziness (Nervous system disorders) | 1/76 | 1/74
Headache (Nervous system disorders) | 1/76 | 6/74
Syncope (Nervous system disorders) | 0/76 | 1/74
Syncope vasovagal (Nervous system disorders) | 0/76 | 2/74
Anxiety (Psychiatric disorders) | 0/76 | 1/74
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0/76 | 1/74
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0/76 | 2/74
Rash (Skin and subcutaneous tissue disorders) | 1/76 | 1/74

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.